CLINICAL TRIAL: NCT02723760
Title: Clinical Study of 99mTc-3PRGD2 SPECT/CT in Diagnosis and Efficacy Evaluation of Rheumatoid Arthritis
Brief Title: 99mTc-3PRGD2 SPECT/CT in Rheumatoid Arthritis Patients
Acronym: TRGDRA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Weibing Miao, PhD, Director, Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAHFMUNM001
Record Dates: First submitted 2016-03-10; First posted 2016-03-30 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 99mTc-3PRGD2 SPECT/CT scanning (Experimental): Determine if 99mTc-3PRGD2 SPECT/CT is safe and effective in diagnosis and efficacy evaluation of rheumatoid arthritis
  Interventions: Drug: 99mTc-3PRGD2

INTERVENTIONS:
Drug: 99mTc-3PRGD2 — SPECT/CT scanning: single intravenous bolus injection of nearly 11.1 MBq/kg body weight of 99mTc-3PRGD2 on rheumatoid arthritis patients, whole-body planar and lesions section for determination the accumulation of 99mTc-3PRGD2 in the joints and other parts of the body.
  For diagnosis study, each patient will be carried out SPECT/CT scanning once. For efficacy evaluation study, each patient will be carried out SPECT/CT scanning three times (before treatment, the midterm treatment and late stage treatment).
  Other Names: 99mTc-HYNIC-3PRGD2

SUMMARY:
This is an open-label SPECT/CT (single photon emission computed tomography/computed tomography) study to investigate the diagnosis and efficacy evaluation performance of 99mTc-3PRGD2 in rheumatoid arthritis patients. A single dose of nearly 11.1 MBq/kg body weight of 99mTc-3PRGD2 (≤20µg 3PRGD2) will be intravenously injected into the patients. Visual and semiquantitative method will be used to assess the whole-body planar and lesions section SPECT/CT images. Adverse events will also be observed in the patients.

DETAILED DESCRIPTION:
As a critical member of adhesion molecule integrin family and an important representative angiogenesis-related molecular, integrin αvβ3 is expressed at low levels on mature endothelial cells and normal cells, but it is overexpressed on the neovasculature endothelial cells, which has a high specificity and affinity in binding to the tri-peptide sequence of arginine-glycine-aspartic acid (RGD). Angiogenesis in the synovial membrane plays an important role in the pathogenesis of rheumatoid arthritis (RA). Therefore, radiolabeled RGD peptides can be used as molecular probe in radionuclide imaging to assess angiogenesis noninvasively in vitro and investigate the progress of RA, so as to achieve the goal of early diagnosis and efficacy evaluation for RA.

Accordingly, a variety of radiolabeled RGD peptides have been used as radiotracers targeting the integrin αvβ3 expression to assess angiogenesis in vitro for noninvasive imaging via PET (positron emission tomography) or SPECT (single photon emission computed tomography). Some radiolabeled cyclic RGD peptides, such as 18F-Galacto-RGD, 18F-AH111585 and 99mTc-NC100692, have been investigated into clinical trials. The results demonstrated that both radiotracers allowed the specific imaging of various types of tumors, and the tumor uptake correlated well with the expression of integrin αvβ3 in both animal models and patients. Recently, several RGD dimeric peptides with PEG linkers have been studied. The new types of RGD peptides showed much higher in vitro integrin αvβ3-binding affinity than the single RGD tri-peptide sequence, and importantly, they exhibited significantly increased tumor uptake and improved in vivo kinetics in animal models. As a representative, 99mTc-3PRGD2 could be easily prepared and exhibited excellent in vivo behaviors in animal models. No adverse reactions are observed in animal models to date.

99mTc-3PRGD2, a novel tracer targeting integrin αvβ3 receptor, was tried to use in some tumors in recent years. However, there are few studies of 99mTc-3PRGD2 in other diseases except for tumors, especially no relevant reports in rheumatoid arthritis. Therefore, the investigators expect to further expand the applications of 99mTc-3PRGD2 in other diseases and to provide new methods and thoughts of assessing the efficacy of anti-αvβ3 or anti-angiogenesis therapy in rheumatoid arthritis. Based on the investigators previous animal study of 99mTc-3PRGD2 in RA, the investigators have strong interests in clinical trials of 99mTc-3PRGD2. An open-label SPECT/CT study has been designed to investigate 99mTc-3PRGD2 SPECT/CT in diagnosis and efficacy evaluation of RA. A single dose of nearly 11.1MBq/kg body weight 99mTc-3PRGD2 (≤20µg 3PRGD2) will be intravenously injected into the patients. Visual and semiquantitative method will be used to assess the whole-body planar and lesions section SPECT/CT images. Adverse events will also be observed in the patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic group:

  * Males and females, ≥20 and ≤ 70 years old.
  * X-ray radiography and/or CT and/or MRI and/or 99mTc-MDP bone scan and/or 18F-FDG PET/CT diagnosis in suspicion of primary or recurrent rheumatoid arthritis (RA).
  * The above patients should be confirmed according to the ACR/EULAR (American rheumatism association and the European Union for resistance rheumatism) diagnostic criteria of RA.
* Efficacy evaluation group:

  * Males and females, ≥20 and ≤ 70 years old.
  * Firstly and definitely diagnose with RA, and prepare to treat.
  * X-ray radiography and/or CT and/or MRI and/or 99mTc-MDP bone scan and/or 18F-FDG PET/CT before treatment, the midterm treatment and late stage treatment (three months after the initial treatment) are available.

Exclusion Criteria:

* Females planning to bear a child recently or with childbearing potential.
* Known severe allergy or hypersensitivity to IV radiographic contrast.
* Inability to lie still for the entire imaging time because of cough, pain, etc.
* Inability to complete the needed examinations due to severe claustrophobia, radiation phobia, etc.
* Concurrent severe and/or uncontrolled and/or unstable other medical disease that, in the opinion of the Investigator, may significantly interfere with study compliance.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
99mTc-3PRGD2 SPECT/CT scan | Two year
  99mTc-3PRGD2 SPECT/CT scan will be carried out in RA patients to implement visual and semiquantitative assessment of arthritic joints. Visual analysis will be performed by consensus reading by at least 3 experienced nuclear medicine physician to observe the the uptake of 99mTc-3PRGD2 on arthritic joints. The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake values (SUVs) of arthritic joints and organs will be measured.

SECONDARY OUTCOMES:
X-ray radiography and/or CT(computed tomograph) and/or MRI(magnetic resonance imaging) | One year
  X-ray radiography and/or CT and/or MRI will be carried out in RA patients to observe the degree of destruction for arthritic joints.
99mTc-MDP bone scan | One year
  99mTc-MDP bone scan will be carried out in RA patients to observe the uptake of arthritic joints and to measure the SUVs of these joints.
18F-FDG PET/CT | One year
  18F-FDG PET/CT will be carried out in RA patients to observe the uptake of arthritic joints and to measure the SUVs of these joints.
Serum rheumatoid factor (RF) | One year
  The patients will be required to test the serum rheumatoid factor routinely.
Serum antinuclear antibodies (ANAs) | One year
  The patients will be required to test the serum antinuclear antibodies routinely.
Erythrocyte sedimentation rate (ESR) | One year
  The patients will be required to test the blood erythrocyte sedimentation rate routinely.
Adverse events collection | 5 days
  Adverse events within 5 days after the injection and scanning of patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, PhD, Study Director — Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Zhu Z, Miao W, Li Q, Dai H, Ma Q, Wang F, Yang A, Jia B, Jing X, Liu S, Shi J, Liu Z, Zhao Z, Wang F, Li F. 99mTc-3PRGD2 for integrin receptor imaging of lung cancer: a multicenter study. J Nucl Med. 2012 May;53(5):716-22. doi: 10.2967/jnumed.111.098988. Epub 2012 Apr 12. PMID 22499615
- [Background] Miao W, Zheng S, Dai H, Wang F, Jin X, Zhu Z, Jia B. Comparison of 99mTc-3PRGD2 integrin receptor imaging with 99mTc-MDP bone scan in diagnosis of bone metastasis in patients with lung cancer: a multicenter study. PLoS One. 2014 Oct 22;9(10):e111221. doi: 10.1371/journal.pone.0111221. eCollection 2014. PMID 25338281
- [Background] Huang C, Zheng Q, Miao W. Study of novel molecular probe 99mTc-3PRGD2 in the diagnosis of rheumatoid arthritis. Nucl Med Commun. 2015 Dec;36(12):1208-14. doi: 10.1097/MNM.0000000000000375. PMID 26352213